CLINICAL TRIAL: NCT00671515
Title: Pioglitazone for the Treatment of Major Depressive Disorder Comorbid With Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph Calabrese, MD (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Joseph Calabrese, MD, Director, Mood Disorders Program, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-07-20
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2016-11

CONDITIONS: Depressive Disorder, Major; Metabolic Syndrome X
Keywords: Depressive Disorder, Major; Metabolic Syndrome X; pioglitazone
MeSH Terms: conditions — Depressive Disorder, Major; Metabolic Syndrome | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pioglitazone (Experimental): An open-label 12-week trial of pioglitazone monotherapy. The investigators will titrate pioglitazone to the maximum tolerable dose up to 45mg per day.
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — An open-label 12-week trial of pioglitazone monotherapy. The investigators will titrate pioglitazone to the maximum tolerable dose up to 45mg per day.
  Other Names: Actos

SUMMARY:
The goal of this study is to begin to test whether or not pioglitazone, an FDA approved medication used to treat high blood sugar, may be safe and effective in treating Major Depressive Disorder (MDD) in patients with comorbid Metabolic Syndrome (METSYN).

ELIGIBILITY:
Inclusion Criteria:

* Be male or female between the ages of 18 and 70
* DSM-IV diagnosis of major depressive disorder
* Currently depressed as confirmed by the MINI-Plus at the screening visit
* Quick Inventory of Depressive Symptomatology-Self-Report(QIDS-SR) score > 11 at study baseline
* Meets criteria for the metabolic syndrome as defined by the NCEP ATP III criteria

Exclusion Criteria:

* Pregnancy or breast feeding
* Unstable or inadequately treated medical illness as judged by the investigator
* Severe personality disorder
* Serious suicidal risk as judged by the investigator or having a score > 2 on item 18 of the Inventory of Depressive Symptomatology-Clinician Rated (IDS-CR) scale
* Known history of intolerance or hypersensitivity to pioglitazone
* Treatment with pioglitazone in the 3 months prior to randomization
* Currently taking an antidiabetic/glucose-lowering agent. Antidiabetic agents that are prohibited include insulin, rosiglitazone, metformin, sitagliptin, sulfonylureas (e.g. glyburide, glipizide, glimepiride), non-sulfonylurea secretagogues (e.g. repaglinide, nateglinide), incretins (e.g. exenatide), and α-glucosidase inhibitors (e.g. acarbose, miglitol).
* Diagnosed with dementia
* Diagnosed with heart failure
* Transaminase elevation >2.5 times the upper limit of normal
* Presence of renal impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-04; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Calabrese, MD, Principal Investigator — University Hospitals Cleveland Medical Center - Mood Disorders Program
Locations (1):
- University Hospitals Cleveland Medical Center - Mood Disorders Program, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Phase 1
Arm/Group | Pioglitazone
Started | 23
Completed | 20
Not Completed | 3
Period: Phase 2
Arm/Group | Pioglitazone
Started | 13
Completed | 9
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Pioglitazone
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (10.2)
Gender [Count of Participants; unit: Participants]
  Female | 20
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Depression Symptom Severity From Baseline to Study Endpoint
Description: Inventory of Depressive Symptoms-Clinician rated, 30 item (IDS-C30) score change from baseline to study endpoint. IDS-C30 total scores can range from 0 to 84, with higher scores indicating a worse outcome
Time Frame: Week 0 - Week 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pioglitazone
Number analyzed (Participants) | 23
Units on a scale | -20.9 (12.1)

2. Secondary Outcome: Change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) From Baseline to Study Endpoint
Description: The homeostatic model assessment (HOMA) is a method used to quantify insulin resistance. Insulin resistance is a condition in which cells fail to respond to the normal actions of the hormone insulin. Typically cutoff of HOMA-IR for identifying those with insulin resistance is 2.5.
Time Frame: Week 0-Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pioglitazone
Number analyzed (Participants) | 23
units on a scale | -0.810 (0.748)

ADVERSE EVENTS:
Arm/Group | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 20/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=23)
Headache (General disorders) | 6 (6)
Dizziness/Lightheadedness (General disorders) | 5 (5)
Increased Appetite (General disorders) | 4 (4)
Weight Gain (General disorders) | 4 (4)
Ankle/Leg Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Blurred Vision (Eye disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Sedation (General disorders) | 2 (2)
Hot Flashes (General disorders) | 2 (2)
Insomnia (General disorders) | 2 (2)
Itching (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes